

Title: A Phase 2, Randomized Study of MLN0128 (a Dual TORC1/2 Inhibitor), MLN0128+MLN1117 (a PI3Kα Inhibitor), Weekly Paclitaxel, or the Combination of Weekly Paclitaxel and MLN0128 in Women With Advanced, Recurrent, or Persistent Endometrial Cancer

NCT Number: NCT02725268

SAP Approve Date: 07 September 2018

Certain information within this Statistical Analysis Plan has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable (PPD) information or company confidential information (CCI).

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.



### STATISTICAL ANALYSIS PLAN

STUDY NUMBER: C31004

the applicable Terms of Use A Phase 2, Randomized Study of MLN0128 (a Dual TQRC1/2 Inhibitor), MLN0128+MLN1117 (a PI3Kα Inhibitor), Weekly Paclitaxel, or the Combination of Weekly Paclitaxel and MLN0128 in Women With Advanced, Recurrent, or Persistent Endometrial Cancer

Version: Final

Date: 07 September 2018

Prepared by:

PPD

Protocol Version: Protocol Am
Protocol Date: 23 January 2018 Protocol Version: Protocol Amendment No. 05

Properly of Takeda: For non-commercial use only and subject to the applicable Terms of use

7.8

| 2.0 | TABLE OF CONTENTS | |
|---|---|---|
| 1.0 | TITLE PAGE | 1 |
| 1. | 1 APPROVAL SIGNATURES | 2 |
| 2.0 | TABLE OF CONTENTS. | 3 |
| 3.0 | LIST OF ABBREVIATIONS | 5 |
| 4.0 | OBJECTIVES | 7 |
| 4. | OBJECTIVES | 7 |
| 4.2 | 2 Secondary Objectives | 7 |
| 4.3 | 3 Quality of Life Objectives | 7 |
| 4.4 | 4 Exploratory Objectives | 7 |
| 4.: | Quality of Life Objectives Exploratory Objectives Study Design 4.5.1 Overview of Study Design ANALYSIS ENDPOINTS Primary Endpoint Secondary Endpoints Quality of Life Endpoints Exploratory Endpoints | 8 |
| | 4.5.1 Overview of Study Design | 8 |
| 5.0 | ANALYSIS ENDPOINTS | 10 |
| 5. | 1 Primary Endpoint | 10 |
| 5.2 | 2 Secondary Endpoints | 10 |
| 5.3 | 3 Quality of Life Endpoints | 10 |
| 5.4 | 4 Exploratory Endpoints | 10 |
| 6.0 | DETERMINATION OF SAMPLE SEE | 12 |
| 7.0 | METHODS OF ANALYSIS AND PRESENTATION | 13 |
| 7. | 1 General Principles | 13 |
| | 7.1.1 Methods for Handling Missing Data | 13 |
| | 7.1.2 Definitions of Baseline Values | |
| | 7.1.3 Definition of Study Days | 14 |
| 7.2 | 2 Analysis Sets | 14 |
| 7.3 | 3 Disposition of Subjects | 15 |
| 7.4 | | |
| 7.: | 5 Medical History and Concurrent Medical Conditions | 16 |
| 7.0 | 6 Medication History and Concomitant Medications | |
| 19 | 7.6.1 Prior Therapies | 17 |
| 4 | 7.6.2 Follow-up Anti-cancer Therapy | 17 |
| O`7. | 7 Study Drug Exposure and Compliance | 17 |
| ) | 7.7.1 Study Treatments | |
| | 7.7.2 Extent of Exposure | 17 |
| | 7.7.3 Action on Drug | 18 |

| 7.8.1 Primary Efficacy Endpoint(s) | 18 |
|---|---|
| 7.8.2 Secondary Efficacy Endpoint(s) | |
| 7.8.3 Additional Efficacy Endpoint(s) | 24 |
| 7.9 Pharmacokinetic/Pharmacodynamic Analysis | <u>(?)</u> 5 |
| 7.9.1 Pharmacokinetic Analysis | 25 |
| 7.9.2 Pharmacodynamic Analysis | 25 |
| 7.9.1 Pharmacokinetic Analysis 7.9.2 Pharmacodynamic Analysis 7.10 Patient Reported Outcomes 7.10.1 EORTC QLQ-C30 and EORTC QLQ-EN24 Scores | 26 |
| 7.10.1 EORTC QLQ-C30 and EORTC QLQ-EN24 Scores | 26 |
| 7.10.2 Percentage of Patients Experiencing Improvement or Deterioration | 26 |
| 7.10.2 T | 20 |
| 7.11 Safety Analysis | 29 |
| 7.11.1 Adverse Events | 29 |
| 7.11.2 Vital Signs | 32 |
| 7.11.3 12-Lead ECGs | 32 |
| 7.11.4 ECOG Performance Status | 33 |
| 7.10.3 Time to Deterioration 7.11 Safety Analysis 7.11.1 Adverse Events 7.11.2 Vital Signs 7.11.3 12-Lead ECGs 7.11.4 ECOG Performance Status 7.12 Interim Analysis 7.13 Changes in the Statistical Analysis Plan | 33 |
| 7.13 Changes in the Statistical Analysis Plan | 34 |
| 8.0 REFERENCES | 35 |
| 9.0 APPENDIX | 36 |
| 9.0 APPENDIX | |

### 3.0 LIST OF ABBREVIATIONS

| C3100<br>Statist | )4<br>tical Analysis Plan | BBREVIATIONS Term adverse event alanine aminotransferase absolute neutrophil count activated partial thromboplastin time aspartate aminotransferase clinical benefit rate complete response case report form computed tomography electrocardiogram Eastern Cooperative Oncology Group electronic case report form electronic data capture European Organization for Research and Treatment of Cancer Quality of Life |
|---|---|---|
| 3.0 | LIST OF AB | BBREVIATIONS |
| Abbre | eviation | Term |
| AE | - | adverse event |
| ALT | | alanine aminotransferase |
| ANC | | absolute neutrophil count |
| aPTT | | activated partial thromboplastin time |
| AST | | aspartate aminotransferase |
| CBR | | clinical benefit rate |
| CR | | complete response |
| CRF | | case report form |
| CT | | computed tomography |
| CCI | 1 | *0 |
| ECG | 1 | electrocardiogram |
| ECOG | ţ | Eastern Cooperative Oncology Group |
| eCRF | | electronic case report form |
| EDC | | electronic data capture |
| | C QLQ-EN24 | European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Endometrial Cancer Module |
| EORT | C QLQ-C30 | European Organization for Research and Treatment of Cancer Quality of Life Questionnaire |
| EOT | | end of treatment |
| INR | | international normalized ratio |
| IRC | | Independent review committee |
| ITT | | intent-to-treat |
| IRT | | Interactive Response Technology |
| MedDI | RA | Medical Dictionary for Regulatory Activities |
| MLN0 | | also known as TAK-228 |
| MRI | | magnetic resonance imaging |
| mTOR | TCAE COLO | mammalian (or mechanistic) target of rapamycin |
| NCI C | TCAE | National Cancer Institute Common Terminology Criteria for Adverse Events |
| ORR | . Y | overall response rate |
| OS | 70. | overall survival |
| PFS | TE. | progression-free survival |
| PI3K | SIL | phosphoinositide 3-kinase |
| PIK3C | <sup>L</sup> A | phosphoinositide-3-kinase, catalytic alpha polypeptide |
| PK | | pharmacokinetic(s) |
| PO | | by mouth (oral) |
| PPI | | proton pump inhibitor |
| PR | | partial response |
| PRO | | patient-reported outcome |
| PTEN | | phosphatase and tensin homolog |
| | | F |

| Abbreviation | Term |
|---|---|
| PT | prothrombin time quaque die; each day; once daily once daily for 3 days each week quality of life rate-corrected QT interval (msec) QT interval (msec) with Fridericia correction once weekly Response Evaluation Criteria in Solid Tumors serious adverse event statistical analysis plan stable disease treatment-emergent adverse events mammalian (or mechanistic) target of rapamycin complex 1 |
| QD | quaque die; each day; once daily |
| QD×3 QW | once daily for 3 days each week |
| QOL | quality of life |
| QTc | rate-corrected QT interval (msec) |
| QTcF | QT interval (msec) with Fridericia correction |
| QW | once weekly |
| RECIST | Response Evaluation Criteria in Solid Tumors |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SD | stable disease |
| TEAE | treatment-emergent adverse events |
| TORC1 | mammalian (or mechanistic) target of rapamycin complex 1 |
| TORC2 | |
| TTP | time to progression upper limit of the normal range white blood cell |
| | upper limit of the normal range |
| WBC | white blood cell |
| | upper limit of the normal range white blood cell |
| perty of Takedai. For | |
| of Co. | |
| certify. | |
| R | |
| 8 | |

### 4.0 OBJECTIVES

### 4.1 Primary Objectives

The primary objective of the study is:

• To determine if MLN0128 in combination with weekly paclitaxel improves progression free survival (PFS) compared to weekly paclitaxel alone.

### 4.2 Secondary Objectives

The secondary objectives of the study are:

- To determine if single-agent MLN0128 improves PFS compared to weekly paclitaxel alone.
- To determine if MLN0128 + MLN1117 improves PFS compared to weekly paclitaxel alone.
- To assess the safety and tolerability of single-agent MLN0128, MLN0128 in combination with paclitaxel, and MLN0128 + MLN1117.
- To evaluate improvement in efficacy measures (endpoints other than PFS) of MLN0128 in combination with weekly paclitaxel, single-agent MLN0128, and MLN0128 + MLN1117 compared to weekly paclitaxel alone.
- To collect plasma concentration-time data with sparse PK sampling to contribute to future population PK analysis.

## 4.3 Quality of Life Objectives

The health-related quality of life (HRQL) objective is:

• To assess the QOL and symptoms in patients treated with MLN0128 in combination with weekly paclitaxel, single-agent MLN0128, and MLN0128 + MLN1117 to weekly paclitaxel alone.

## 4.4 Exploratory Objectives

The exploratory objectives of the study are:

### 4.5 Study Design

### 4.5.1 Overview of Study Design

This study is a phase 2, open-label, randomized, multicenter, 4-arm study of the safety and efficacy of MLN0128 in combination with paclitaxel, single-agent MLN0128, single-agent paclitaxel, and MLN0128 in combination with MLN1117 in adult women with advanced endometrial cancer. The patient population will consist of women with histologic or cytologic diagnosis of endometrial carcinoma (including endometrioid, serous, mixed adenocarcinoma, clear-cell carcinoma, or carcinosarcoma) that is advanced, recurrent, or persistent, that has relapsed or is refractory to curative therapy or established treatments. Patients must have had 1 prior platinum-based chemotherapeutic regimen, but not more than 2 prior systemic chemotherapy regimens.

Eligibility will be determined during the Screening period, which may last for up to 28 days before the Cycle 1, Day 1 visit. Patients who meet all eligibility criteria and provide written informed consent will be enrolled in this study. Study drug will be administered in 28-day treatment cycles.

Approximately 242 patients will be randomized at a ratio of 1:1:1:1 to receive study drug in 1 of 4 treatment arms:

Arm A: paclitaxel 80 mg/m2 weekly on Days 1, 8, and 15 of a 28-day cycle

Arm B: paclitaxel 80 mg/m2 weekly on Days 1, 8, and 15 of a 28-day cycle

+ MLN0128 4 mg on Days 2-4, 9-11, 16-18, and 23-25 of a 28-day cycle

Arm C: MLN0128 30 mg once weekly (QW) on Days 1, 8, 15, and 22 of a 28-day cycle

Arm D: MLN0128 4 mg + MLN1117 200 mg on Days 1-3, 8-10, 15-17, and 22-24 of a 28-day cycle

A centralized randomization will be used with the following stratification factors:

- Histological subtype: endometrioid vs. nonendometrioid.
- Lines(s) of prior chemotherapy: 1 vs. 2.
- Prior taxane therapy (other than weekly): yes vs. no.

In the event that enrollment into a treatment arm(s) is closed, patients will be randomized 1:1 into the remaining treatment arms. Paclitaxel will be administered intravenously (IV) while MLN0128 and MLN1117 will be administered PO throughout the study. Patients in Arm A and Arm B will receive paclitaxel alone or paclitaxel + MLN0128 until they experience disease progression, unacceptable toxicity, or withdraw consent. Patients in Arm B who discontinue paclitaxel prior to disease progression may continue to receive MLN0128 alone until they experience disease progression, unacceptable toxicity, or withdraw consent. In addition, patients will receive MLN0128 (in Arm C) or MLN0128 + MLN1117 (in Arm D) continuously until they experience disease progression, unacceptable toxicity, or withdraw consent. Patients who

discontinue study treatment for reasons other than progressive disease will continue to have PFS follow-up visits every 2 months ( $\pm$  1 week) for the first 6 months after the end-of-treatment (EOT) visit, then every 3 months ( $\pm$  1 week) until disease progression, death, or start of another anticancer therapy, whichever occurs first. After disease progression, patients will be followed for OS every 3 months ( $\pm$  1 week).

Patients will attend the EOT visit 30 to 40 days after receiving their last dose of study drug.

Sparse PK samples will be collected from patients enrolled in Arms B, C, and D for determination of the plasma concentration of MLN0128 and/or MLN1117 during Cycle 1 at prespecified time points as described in the Pharmacokinetic Sample Breakdown table in the study protocol. Data generated in this study will be combined with data from other studies in which the PK of MLN0128 is characterized for population PK analysis. For correlative biomarker analysis, fresh and archival tumor samples will be obtained during screening, as well as a blood sample for at prespecified time points as described in the Schedule of Events in the study protocol. In addition, fresh tumor samples will be obtained 2 to 4 hours after dosing on Cycle 1 Day 22 from patients in Arms C and D to identify adaptive response mechanisms to treatment of MLN0128 or MLN0128 + MLN1117.

Radiological tumor evaluations (computed tomography [CT] scan with IV contrast or magnetic resonance imaging [MRI], as clinically indicated) of the chest, abdomen, and pelvis will be used to evaluate disease response according to Response Evaluation Criteria in Solid Tumors (RECIST) guidelines (Version 1.1). Radiographic tumor evaluations will be performed at the time points specified in the Schedule of Events in the study protocol.

Changes in QOL disease-specific symptoms will be assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) and the Endometrial Cancer Module (EORTC QLQ-EN24). In addition to assessing selected symptoms, these instruments will measure the effects of disease and treatment on physical, role, emotional, cognitive, and social functioning.

Toxicity will be evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 4.03, effective date 14 June 2010.

Adverse events will be assessed, and laboratory values, vital signs, and electrocardiograms will be obtained to evaluate the safety and tolerability of MLN0128 in combination with paclitaxel, single-agent MLN0128, and MLN0128 + MLN1117.

There will be 2 interim analyses with early stopping rules for futility in the single-agent MLN0128 arm (Arm C) and MLN0128+MLN1117 arm (Arm D).

### 5.0 ANALYSIS ENDPOINTS

### 5.1 Primary Endpoint

The primary endpoint is Progression Free Survival (PFS).

### 5.2 Secondary Endpoints

The secondary endpoints are:

- The number and percentage of patients with treatment-emergent adverse events (TEAEs).
- Overall survival (OS).
- Time-to-progression (TTP).
- Objective response rate (ORR; defined as complete response [CR]+partial response [PR] per Response Evaluation Criteria in Solid Tumors [RECIST] Version 1.1).
- Clinical benefit rate (CBR; defined as CR+PR+stable disease (SD)) with SD of any duration.
- CBR at 16 weeks (CBR-16 is defined as the proportion of patients who achieve CR or PR of any duration or have SD with a duration of at least 16 weeks).

### 5.3 Quality of Life Endpoints

The QOL endpoints are:

- Change from baseline in the EORTCQLQ-C30 global health status (GHS)/QOL score to end of study visit.
- Change from baseline in the EORTC QLQ-C30 functioning score to end of study visit.
- Change from baseline in the EORTC QLQ-C30 symptom score to end of study visit.
- Change from baseline in the EORTC QLQ-EN24 score to the end of study visit.

## 5.4 Exploratory Endpoints

The exploratory endpoints are:



Properly of Takeda: For non-commercial use only and subject to the applicable Terms of use

Ine primary efficacy endpoint of the study is PFS and the primary comparison is between the paclitaxel and the paclitaxel + MLN0128 4 mg QDx3 treatment arm. Assuming the median PFS is 4 months for paclitaxel and paclitaxel + MLN0128 4 mg QDx3 can improve the median to 6.5 months (hazard ratio of 0.615, approximately 38% reduction in the hazard rate) a total of 124 PFS events and 90 patients per treatment arm are required. The call of 80%, 2-sided alpha of 5% and a light of 124 per call of consent. Enrollment to the third treatment arm of single-agent MLN0128 30 mg QW and the fourth treatment arm of MLN0128 4 mg QDx3 in combination with 200 mg MLN1117 has been closed. The total sample size for the study will be approximately 242 patients.

The total accrual duration will be approximately 25 months to complete enrollment in the ent am months aft monte on marconing relative only and sulfill and paclitaxel and paclitaxel+MLN0128 4 mg QD×3 treatment arms. The final analysis for the primary comparison of PFS between the paclitaxel treatment arm and the paclitaxel + MLN0128 4 mg QDx3 treatment arm will occur approximately 5 months after the last patient is

### 7.0 METHODS OF ANALYSIS AND PRESENTATION

### 7.1 General Principles

All statistical analyses will be conducted using SAS® Version 9.4.

Continuous data will be summarized using descriptive statistics (number of observations, mean, standard deviation, median, 25<sup>th</sup> and 75<sup>th</sup> percentiles (where specified), minimum, and maximum). Frequencies and percentages will be used for summarizing categorical (discrete) data. For summaries of categorical variables percentages are based on the number of subjects with non-missing values unless otherwise specified (e.g. objective response rate, clinical benefit rate, CBR at 16 weeks).

Confidence intervals, when presented, will generally be constructed at the 95% level. For binomial variables, the normal approximation methods will be employed unless otherwise specified.

All statistical tests and resulting p-values will be reported as 2-sided and will be assessed at  $\alpha$ =0.05 significance level unless otherwise stated. P-values should be presented to 3 decimal places, with values less than 0.001 presented as <0.001.

Means and medians will be presented to 1 more decimal place than the recorded data. The standard deviations (SDs) will be presented to 2 more decimal places than the recorded data. Confidence intervals about a parameter estimate will be presented using the same number of decimal places as the parameter estimate. Percentages will be presented to 1 decimal place.

A month is operationally defined to be 30.4375 days.

Where specified, there will be three pair-wise comparisons between paclitaxel vs. paclitaxel+MLN0128, between paclitaxel vs. MLN0128 and between paclitaxel vs. MLN0128+MLN1117.

## 7.1.1 Methods for Handling Missing Data

For efficacy and safety data, no imputation of values for missing data will be performed. For patient reported outcomes, handling of missing data is discussed in section 7.10. Data imputation rules for incomplete dates are described in Appendix B.

## 7.1.2 Definitions of Baseline Values

In general, for efficacy endpoints the last observed measurement prior to randomization will be considered the baseline measurement. For safety end points the last observation before first dose of study drug will be considered the baseline measurement. For patient-reported outcomes the last observed measurement on or before the date of first dose of study drug will be considered the baseline measurement.

### 7.1.3 Definition of Study Days

For the purpose of efficacy data summary, Day 1 is defined as the date of randomization. For visits (or events) that occur on or after randomization, Day is defined as (date of visit [event] – date of randomization + 1). For visits (or events) that occur prior to randomization, Day is defined as (date of visit [event] – date of randomization). There is no Day 0.

For the purpose of safety data summary or calculations of time since baseline, Study Day 1 is defined as the date on which a subject is administered their first dose of study drug. For visits (or events) that occur on or after the first dose of study drug, study day is defined as (date of visit [event] – date of first dose of study drug + 1). For visits (or events) that occur prior to Study Day 1, study day is defined as (date of visit [event] – date of first dose of study drug). There is no Study Day 0.

### 7.2 Analysis Sets

- Intent-to-treat (ITT) population: all randomized patients. Patients will be analyzed according to the randomization assignment. The ITT population will be used for the primary efficacy analysis of PFS, and secondary efficacy endpoints including OS and TTP.
- Safety population: patients who receive at least 1 dose of study drug. Patients will be analyzed according to the treatment arm actually received. The safety population will be used for all safety analyses. In addition, the safety population will be used for a sensitivity analysis of secondary efficacy endpoints ORR, CBR and CBR-16 and the best overall response and patients will be analyzed according to the randomization assignment.
- Response-evaluable population: patients who receive at least 1 dose of study drug, have measurable disease at Baseline, and have 1 post-Baseline disease assessment. Patients will be analyzed according to the randomization assignment. The response-evaluable population will be used for the primary analysis of secondary efficacy endpoints of ORR, CBR and CBR-16, and the best overall response.
- Per-protocol population: all ITT patients who meet the following criteria:
  - Had at least one adequate post-randomization tumor assessment.
  - Received treatment as randomized.
  - Did not have any major or important protocol deviations that would potentially impact the interpretation of the efficacy analyses.

The subset of major/important protocol deviations that would exclude a patient from the per protocol population will be based on a review of the protocol deviations in the clinical trial management system and will be documented prior to database lock. The perprotocol population will be used for a sensitivity analysis of PFS, and secondary efficacy endpoints including OS and TTP.

The number and percentage of patients in each population will be summarized.

### 7.3 **Disposition of Subjects**

Study information including the date first subject signed ICF, date of last subject's last visit/contact, date of last subject's last procedure for collection of data for primary endpoint of PFS, MedDRA version, WHO Drug version and SAS Version will be generated in a summary table. The date of last procedure for PFS is the date of progressive disease or death, otherwise use the date of the last response assessment.

The disposition of patients includes the number and percentage of patients for the following categories: randomized and not treated, discontinued study drug, primary reason to discontinue study drug, ongoing (if applicable at the time of DB lock), discontinued from the study, and primary reason to discontinue from the study. All percentages will be based on the number of patients in the ITT population.

### 7.4 **Demographic and Other Baseline Characteristics**

ialuse only and sul Summaries of demographics, baseline characteristics and stratification factors will be presented for subjects in the ITT population.

The demographic characteristics consist of:

- Age (continuous)
- Age category 1
  - $\circ$  < 65 years
  - $\circ \geq 65 \text{ years}$
- Age category 2
  - Adults (18-64 years
  - o From 65 to 84 years
  - o 85 years and over
- Height (cm)
- Weight (kg) screening if available otherwise C1D1
- Ethnicity
- Race
- Geographic Region, Country, Site

Australia and New Zealand

North America

- Canada
- United States

### Europe

- Belgium
- Germany
- Italy
- Netherlands
- Norway
- Spain
- United Kingdom

### Baseline characteristics consist of:

- Time since initial diagnosis (months) [date of first dose date of initial diagnosis/(30.4375))].
- Histological classification [Endometrioid adenocarcinoma, NOS; Serous cystadenocarcinoma, NOS; Mixed cell adenocarcinoma; Clear cell adenocarcinoma, NOS; Carcinosarcoma, NOS; Unknown].
- Histological grade [Well differentiated (G1); Moderately differentiated (G2); Poorly differentiated (G3); Undifferentiated (G4)].
- ER status
- PR status
- Microsatellite stability
- ECOG Performance Status (categorical)

# Stratification factors consist of:

- Histological subtype: endometrioid vs. non-endometrioid
- Prior lines of chemotherapy: 1 vs. 2
- Prior taxane therapy: yes vs. no.

There will be separate summaries for stratification by original IRT and corrected IRT.

## 7.5 Medical History and Concurrent Medical Conditions

No summary for medical history and concurrent medical conditions.

### 7.6 Medication History and Concomitant Medications

No summary for medication history.

The number and percentage of patients taking concomitant medications will be tabulated by WHO standardized medication name based on safety population. Concomitant medications are

medications ongoing at the time of the first dose of study drug or medications that started after first dose and within 30 days of the last dose of study drug.

### 7.6.1 Prior Therapies

The number and percentage of patients with prior radiation, and prior anti-cancer therapies will be summarized based on safety population. The following will be summarized for those patients with prior anti-cancer therapies:

- Type of prior anti-cancer therapy (WHO drug standardized medication name). ine ale
- Best response to most recent prior therapy.
- Prior therapy in the adjuvant setting (Y, N).
- First systemic chemotherapy for metastatic disease (Y, N).

### 7.6.2 Follow-up Anti-cancer Therapy

Number and percentage of patients receiving any anti-cancer therapy, and type of anti-cancer therapy will be summarized based on safety population.

### Study Drug Exposure and Compliance 7.7

### 7.7.1 **Study Treatments**

Cycles consist of 28 days for all treatment arms. In Treatment Arm A, paclitaxel will be administered weekly on Days 1, 8, 15 of a 28-day cycle. In Treatment Arm B, paclitaxel will be administered weekly on Days 1, 8, 15 of a 28-day cycle + MLN0128 administered on Days 2-4, 9-11, 16-18 and 23-25 of a 28-day cycle. In Treatment Arm C, MLN0128 will be administered once weekly on Days 1, 8, 15, and 22 of a 28-day cycle. In Treatment Arm D, MLN0128 and MLN1117 will be administered together, 3 consecutive days per week (on Days 1-3, 8-10, 15-17, and 22-24 of a 28-day treatment cycle), and should be taken on the same days of each week.

### **Extent of Exposure** 7.7.2

Summaries and descriptive statistics of duration of treatment in weeks ((last dose date – start dose date  $\pm \sqrt{3}$ , total number of cycles administered, cumulative dose for each study drug, planned cumulative dose for each study drug and relative dose intensity will be summarized by treatment arm for patients in the safety population. For patients who discontinued Paclitaxel but stayed on MLN0128, number of treatment cycles will be summarized.

Number of cycles administered = A treated cycle is defined as a cycle in which the patient received any amount of study drug. This is defined as Actual Dose greater than zero for at least one of the dosing day in the cycle for any study drug.

Cumulative dose (mg) = Sum of all doses (mg) administered to a subject during the treatment period.

Relative dose intensity = cumulative dose / planned cumulative dose.

Cumulative dose (mg) / [Number of planned dose from start dose date to last dose date\*80mg/m²] \* 100

Number of planned dose = Number of completed 28 documents doses per cycle + Number of cycl

### MLN0128 QDx3 (Days 2-4, 9-11, 16-18 and 23-25 of a 28-day cycle)

### MLN1117 / MLN0128 (Days 1-3, 8-10, 15-17 and 22-24 of a 28-day cycle)

Relative dose intensity (%) presented separately for MLN0128 and MLN1117 is defined as:

{Cumulative dose (mg) / [Number of planned dose from start dose date to last dose date\*Starting dose]} \* 100

Number of planned dose = Number of completed week from start dose date to last dose date\*3 doses per week + Number of doses in the uncompleted week

## MLN0128 QW (Days 1, 8, 15 and 22 of a 28-day cycle)

Relative dose intensity for MLN0128 (%) is defined as:

Cumulative dose (mg) / [Number of planned dose from start dose date to last dose date\*30mg] \* 100

Number of planned dose = Number of completed 28-day cycle from start dose date to last dose date\*4 doses per cycle + Number of doses in the uncompleted cycle

### 7.7.3 Action on Drug

Action on study drug will be summarized by each cycle (Cycles 1-8) and total, for each treatment arm in the safety population.

### **Efficacy Analysis** 7.8

The analysis of PFS, OS and TTP will be based on the ITT population and the PP population. The analysis of ORR, CBR and CBR-16 will be based on both safety and response-evaluable analysis populations. The primary analysis for all efficacy endpoints are based on the investigator response assessment per RECIST 1.1 criteria.

# 7.8.1 Primary Efficacy Endpoint(s)

The primary endpoint is PFS, defined as the time from the date of randomization to the date of first documentation of progression or death due to any cause, whichever occurs first. Progression is based on the investigator response assessment per RECIST 1.1 criteria. PFS in months is defined as:

PFS (months) = (earliest date of progression or death – date of randomization + 1)/30.4375

In the event of progression, the date of progression is defined as the earliest date among target lesions, non-target and new lesions dates at that particular visit.

For a patient whose disease has not progressed and is last known to be alive, PFS will be censored at the last response assessment that is SD or better.

The approach for handling of missing response assessments and censoring is presented in Table 7.a.

Table 7.a Handling of Missing Response Assessment and Censoring ?

| Situation | Date of Progression or<br>Censoring | Outcome |
|---|---|---|
| No baseline tumor assessment | Randomization | Censored |
| No post baseline tumor assessment and no death | Randomization | Censored |
| Disease progression<br>documented between<br>scheduled visits | Date of first documented disease progression | Progressed |
| Disease progression<br>documented subsequent to<br>missing 2 or more adequate<br>tumor assessments | Date of first documented disease progression | Progressed |
| No documented disease progression or no death | Date of last adequate assessment | Censored |
| Alternate subsequent therapy started prior to disease progression | Date of last adequate assessment prior to the start of subsequent therapy | Censored |
| Death without progression and without subsequent anti-<br>cancer therapy | Date of death | Progressed |

# **Adequate Assessments**

Functionally this corresponds to a response assessment with an investigator's assessment other than not evaluable or missing (i.e. CR, PR, SD or PD).

### **PFS Analysis**

The primary efficacy analysis will be based on the ITT population. The Kaplan-Meier method will be used to analyze the distribution of PFS for each treatment arm. Kaplan-Meier survival curves, the 25th, 50th (median), and 75th percentiles, along with associated 2-sided 95% confidence intervals (CIs) based on Brookmeyer and Crowley, and Kaplan-Meier estimates with 95% CIs at 6, 12 and 18 and 24 months will be presented. The primary hypothesis will be tested at the 0.1 significance level (1-sided). The p-values from a stratified log-rank test and hazard ratios (and 95% CI) estimated from a stratified Cox regression model with treatment arm and stratification factors as covariates will be presented for comparison of paclitaxel to paclitaxel+MLN0128, paclitaxel to MLN0128 and paclitaxel to MLN0128+MLN1117. The stratification factors are the histological subtype (endometrioid vs. non-endometrioid), the lines of prior chemotherapy (1vs. 2) and prior taxane therapy (yes vs. no). The original IRT stratification factors will be used in models.

The source of PFS (death or progressive disease) will be summarized by treatment group.

The reasons for censoring in the PFS Kaplan-Meier analysis will be tabulated for each treatment group:

- Received subsequent anti-cancer therapy.
- No baseline or no post baseline response assessment.
- Death or progression after more than 1 missed visit.
- Withdrawal of consent.
- Lost to follow-up.
- No documented death or disease progression.

## 7.8.1.1 Sensitivity Analyses of the Primary Efficacy Endpoint (PFS)

Sensitivity analyses will be performed in order to explore the robustness of the results of the primary analysis.

# PFS Sensitivity Analysis 1: account for missing tumor assessment prior to PFS event (progression or death).

This analysis will be performed only if at least 20% of events of disease progression were documented subsequent to missing 2 or more adequate tumor assessments.

- Subjects who miss 2 or more consecutive adequate scheduled tumor assessments immediately followed by an event of disease progression will be censored on the date of their most-recent adequate tumor assessment prior to the missing/inadequate assessments.
- If 2 or more consecutive missing adequate assessments are immediately followed by an adequate assessment with an overall response assignment of SD, PR, or CR, this will deemed sufficient clinical evidence that progression did not occur during the period of missing data and the missing evaluations will be ignored.

# PFS Sensitivity Analysis 2: discrepancy between original stratification in IRT system and corrected stratification in IRT system

The p-values from a stratified log rank test and the hazard ratio along with its 95% confidence interval will be estimated using a stratified Cox regression model with treatment arm and stratification factors as covariates. PFS will be compared between treatment groups using the corrected IRT strata. This analysis will be performed if at least one stratification variable between the original IRT and the corrected IRT disagrees for at least 10% of the randomized subjects.

# PFS Sensitivity Analysis 3: repeat the primary PFS analysis using the per-protocol population

PFS Sensitivity Analysis 4: repeat the primary PFS analysis based on IRC assessment (see section 7.8.3)

### 7.8.1.2 Subgroup Analyses

The analysis of PFS will be repeated in each of the following subgroups. The focus of the subgroup analyses is to assess the consistency of treatment effects and to present number of patients with events/censored, 25<sup>th</sup>, median and 75<sup>th</sup> percentile with HR and 95% CI within each subgroup for the 3 comparisons: paclitaxel vs. paclitaxel+MLN0128, paclitaxel vs. MLN0128 and paclitaxel vs. MLN0128+MLN1117. In addition, number of events/number of patients, HR and 95% CI within each subgroup for the 3 treatment comparisons will be presented as part of the forest plots and individual Kaplan-Meier survival curves for each subgroup will be presented.

- Age (< 65 years,  $\ge 65$  years).
- Race (white, non-White) [Not Reported will be excluded].
- Region (North America, outside of North America).

Stratification factors per IRT (original):

- Histological subtype (endometrioid vs. non-endometrioid).
- Lines of prior chemotherapy (1 vs. 2).
- Prior taxane therapy (yes vs. no).

# 7.8.2 Secondary Efficacy Endpoint(s)

Secondary efficacy endpoints include OS, ORR, TTP, CBR with SD of any duration, and CBR with SD duration of at least 16 weeks. The analyses of OS and TTP will be done for both the ITT and the per-protocol populations. The analyses of ORR, CBR and CBR-16 will be done for both the safety and response-evaluable populations.

In the event of response (i.e. overall response is PR or better), the date used for start of response is defined as the latest of all dates among target lesions or non-target lesions dates at that particular visit.

### Overall survival (OS)

Overall survival in months is defined as the time from the date of randomization to the date of death [date of death (OS (months) = (date of death – date of randomization + 1)/30.4375)]. Patients without documentation of death at the time of analysis will be censored at the date last known to be alive. The Kaplan-Meier method will be used to analyze the distribution of OS for each treatment arm. Kaplan-Meier survival curves, the 25th, 50th (median), and 75th percentiles, along with associated 2-sided 95% confidence intervals (CIs), and Kaplan-Meier estimates with 95% CIs at 6, 12 and 18 and 24 months will be presented. A stratified log-rank test and hazard ratios (and 95% CI) estimated from a stratified Cox regression model with treatment arm and stratification factors as covariates will be presented for comparison of paclitaxel to paclitaxel+MLN0128, paclitaxel to MLN0128 and paclitaxel to MLN0128+MLN1117. The stratification factors are the histological subtype (endometrioid vs. non-endometrioid), the lines of prior chemotherapy (1vs. 2) and prior taxane therapy (yes vs. no). The original IRT stratification factors will be used in models.

### **Best Overall Response**

Best overall response is defined as the best response recorded after the first dose of study drug until subsequent therapy.

Best Overall Response (unconfirmed): This will be the best response reported by the investigator; ordered from best to worst: Complete Response, Partial Response, Stable Disease, Progressive Disease. The best response can also be Not Evaluable (NE) or No assessment performed if this is the only investigator assessment of objective response available for the patient.

Best Overall Response (confirmed): This will be the best response reported by the investigator; ordered from best to worst: Complete Response, Partial Response, Stable Disease, Progressive Disease. Complete or partial responses may be claimed as best response only if the criteria for each are met at a subsequent time. For the best overall response (confirmed), the confirmation derivation rules will be as described in the following table.

| Overall response 1 <sup>st</sup> time point | Overall response subsequent time point | BEST overall response |
|---|---|---|
| CR C | CR | CR |
| CR | PR | PR |
| CR | SD | SD |
| CR C | PD | SD |
| CR | NE | SD |
| PR | CR | PR |
| PR | PR | PR |
| PR | SD | SD |
| PR | PD | SD |
| PR | NE | SD |
| NE | NE | NE |

Note: No adjustment for a minimum criteria for SD is needed as the first protocol scan is at the end of cycle 2, approximately 8 weeks from first dose.

Overall response rate (ORR) is defined as the proportion of patients among response evaluable population who achieve a best overall response of CR or PR based on investigators assessment of response following RECIST 1.1. ORR will be summarized by both ORR based on unconfirmed best response and ORR based on confirmed best response. A stratified Cochran-Mantel-Haenszel (CMH) test based on stratification factors will be used to compare ORR between treatment arms based on the original IRT (paclitaxel vs. paclitaxel+MLN0128, paclitaxel vs. MLN0128 and paclitaxel vs. MLN0128+MLN1117). The Mantel-Haenszel estimate of the odds ratio and the associated 95% CIs will be presented for each comparison specified above based on original IRT.

### **Clinical Benefit Rate (CBR)**

CBR is defined as the proportion of patients who achieve a best response of CR, PR, or SD of any duration. CBR will be presented for both CBR based on unconfirmed best response and CBR based on confirmed best response. A stratified Cochran-Mantel-Haenszel (CMH) test based on stratification factors will be used to compare CBR between treatment arms (paclitaxel vs. paclitaxel+MLN0128, paclitaxel vs. MLN0128 and paclitaxel vs. MLN0128+MLN1117). The Mantel-Haenszel estimate of the odds ratio and the associated 95% CIs will be presented for each comparison specified above.

### Clinical Benefit Rate at 16 weeks (CBR-16)

CBR at 16 weeks (CBR-16) is defined as the proportion of patients who achieve CR or PR of any duration or have SD with a duration of at least 16 weeks (see below). CBR-16 will be summarized based on unconfirmed best response and confirmed best response. A stratified Cochran-Mantel-Haenszel (CMH) test based on stratification factors will be used to compare CBR-16 between treatment arms (paclitaxel vs. paclitaxel+MLN0128, paclitaxel vs. MLN0128 and paclitaxel vs. MLN0128+MLN1117). The Mantel-Haenszel estimate of the odds ratio and the associated 95% CIs will be presented for each comparison specified above.

SD for at least 16 weeks is a subset of SD, only calculated for those patients with a best response of SD. It is defined as SD at the end of Cycle 2 and at the end of Cycle 4 (see below for exceptions).

CBR at 16 weeks (unconfirmed) is defined as the number of patients who achieve CR or PR at any time or have SD for at least 16 weeks (at the end of Cycle 2 and at the end of Cycle 4).

CBR at 16 weeks (confirmed) is defined as the number of patients who achieve confirmed CR or confirmed PR at any time or have SD for at least 16 weeks or meet the following criteria:

| Overall response at end of Cycle 2 | Overall response at end of Cycle 4 | Meet criteria for SD for at least 16 weeks? |
|---|---|---|
| CR/PR (unconfirmed) | SD | YES |
| SD | CR/PR (unconfirmed) | YES |

In addition, the proportion of patients in the following categories will be summarized by treatment group: CR, PR, SD, SD at least 16 weeks, overall response (ORR), CBR and CBR-16 weeks.

### **Time to Tumor Progression (TTP)**

TTP in months is defined as the time from the date of randomization to the date of first documentation of progression [ (date of first documentation of progression – date of randomization + 1)/30.4375)]. For a patient whose disease has not progressed, TTP will be censored at the last response assessment that is SD or better.

The Kaplan-Meier method will be used to analyze the distribution of TTP for each treatment arm. Kaplan-Meier survival curves, the 25th, 50th (median), and 75th percentiles, along with associated 2-sided 95% confidence intervals (CIs), and Kaplan-Meier estimates with 95% CIs at 6, 12 and 18 and 24 months will be presented. A stratified log-rank test and hazard ratios (and 95% CI) estimated from a stratified Cox regression model with treatment arm and stratification factors as covariates will be presented for comparison of paclitaxel to paclitaxel+MLN0128, paclitaxel to MLN0128 and paclitaxel to MLN0128+MLN1117. The stratification factors are the histological subtype (endometrioid vs. non-endometrioid), the lines of prior chemotherapy (1vs. 2) and prior taxane therapy (yes vs. no). The original IRT stratification factors will be used in models.

### 7.8.3 Additional Efficacy Endpoint(s)

The duration of objective response (DOR) will be calculated for those patients with a best response of CR or PR (for both unconfirmed and confirmed), and is defined as the number of days from the start date of CR, or PR (whichever response is achieved first) until progressive disease or until the last adequate response assessment if there is no progressive disease. The analysis of duration of response will be descriptive in nature and will be based on response-evaluable population.

Waterfall plots of the best percentage change from baseline in the sum of the longest diameter (SLD) of the target lesions will be generated for each treatment group using the response-evaluable population. If one of the target lesion measurements is missing at a visit then the SLD at that visit will not be used for selecting the best percentage change from baseline in SLD for the waterfall plot. The sum of longest diameters (SLD) will be calculated based on the following rules:

- 1. If a target lesion at a visit is "too small to measure", per the CRF completion guidelines the value of 5 mm should have been entered as the diameter. This would be used to calculate the SLD.
- 2. If 2 target lesions conjoin into a single lesion (status="coalesce"), per the CRF completion guidelines the LD of the resulting merged lesion is divided by 2 and reported in the CRF for each of the previous TL and then would be included in the SLD.
- 3. If a target lesion splits into 2 lesions (status="split"), the LDs of the fragmented portions are added up and reported in the CRF and would be included in the SLD.
- 4. Sum of the target lesions (SLD) [in mm] is defined as the sum of the longest diameters of all target lesions at each visit.

- SLD at visit x" "SLD at baseline". Baseline SLD

  corresponds to the SLD from the screening visit.

  6. Percentage change from baseline in SLD [in %] is defined as "SLD change from baseline at visit x" / "SLD at baseline" \* 100.

  7. Best percentage change in SLD is defined as the percentage the visit with the smallest SLD \*\*\*

  All :

All images will be collected and quality controlled by a sponsor-specified central imaging vendor. The independent review committee (IRC) will consist of two independent readers, and an adjudicator. For analysis purposes, if the response assessment at a specific timepoint differs between the 2 readers, the adjudicated response assessment will be used.

The concordance in the assessment of progressive disease between the investigator (INV) and the IRC will be summarized for the ITT population for Arms A (paclitaxel) and B (paclitaxel + MLN0128):

- Agreement on PD status
  - o PD by both IRC and investigator
    - IRC and investigator agree on timing
    - IRC earlier than investigator
    - IRC later than investigator
  - No PD by either IRC or Investigator
- Disagreement on PD status
  - PD by Investigator but not by IRC
  - o PD by IRC but not by investigator

Sensitivity analyses for time-to-event endpoints (PFS, TTP) based on the ITT population and response endpoints (ORR and CBR both unconfirmed and confirmed) for the safety population will be generated based on results from the IRC for Arms A (paclitaxel) and B (paclitaxel + MLN0128).

### 7.9 Pharmacokinetic/Pharmacodynamic Analysis

### Pharmacokinetic Analysis 7.9.1

Sparse PK data for MLN0128 and MLN1117 are being collected to contribute to a future population PK analysis. These data may be combined with data from other studies in which the PK of MLN0128 or MLN1117 is characterized for population PK analysis. The results of population PK analysis will be presented in a separate report.

### Pharmacodynamic Analysis

Biomarker analyses will be exploratory in nature and will be summarized in a separate report.

auent-reported outcome (PRO) assessments will be collected through 2 different instruments: EORTC QLQ-C30 and EORTC QLQ-EN24. The ITT population will be used to present patient reported outcome analysis. For each treatment group and at each assessment point and overall will be summarized. Compliance is defend to the EORTC OLQ-C30 and T30 will be summarized. Compliance is defend to (answered at least one question) as a proportion of the number of expected questionnaires per the schedule of events (Day 1 of each cycle and End of Treatment). Patients who died will not be included in the expected count.

Patient with missing baseline scores are not assessable for baseline description or change from baseline and time to deterioration analyses. Patients with baseline scores, but with no follow-up scores, are not assessable for change from baseline. For time to deterioration they will be censored at Day 1. Published manuals/guidance for EORTC OLO-C30 will be used for scoring and handling missing data. In the case where there is no guidance for handling missing data, missing items will be considered missing, they will not be imputed.

### 7.10.1 EORTC QLQ-C30 and EORTC QLQ-EN24 Scores

Descriptive statistics including the 95% CI around mean for actual values and the change from baseline (post – baseline) will be tabulated at each scheduled time point and the EOT visit for each of the functional and symptom scores from the EORTC QLQ-C30 and QLQ-EN24 questionnaires, the global health status/QOL score and summary score from the EORTC QLQ-C30 questionnaire up to 12 cycles. In addition, the mean and mean change from baseline of the EORTC QLQ-C30 subscales, the global health status/QOL score, summary score and the EORTC QLQ-EN24 subscales will also be presented over time by treatment group in figures up to 12 cycles (including 95% CI around mean).

The change from baseline of EORTC QLQ-C30 subscales, global health status/QOL, summary score and EORTC QLQ-EN24 subscales will be analyzed using linear mixed models, including treatment group, visit, the interaction between treatment group and visit, baseline score (and other covariates i.e. stratification factors as per original IRT) as covariates. Random-intercept only model with appropriate covariance structure will be used based on the following covariance structure in order from unstructured, spatial-power and AR(1). The first covariance structure that has all the parameter estimates converged for all the subscales will be used. The estimated means with 95% CIs will be provided at each time point up to 12 cycles for each treatment arm. The mean differences in each score and 95% CIs and p values for the pairwise comparison of paclitaxel to paclitaxel+MLN0128, paclitaxel to MLN0128 and paclitaxel to MLN0128+MLN1117 will be presented at each time point up to 12 cycles.

### 7.10.2 Percentage of Patients Experiencing Improvement or Deterioration

The subscale scores based on EORTC QLQ-C30 and EORTC QLQ-EN24 and corresponding minimally important differences (MIDs) are defined as shown in Table 7.2. For EORTC QLQ- EN24, the MID threshold of 5 is used in the absence of referenced MID, which corresponded to the value found in the literature for the other scales of the EORTC questionnaire.

Table 7.b Definition of Minimally Important Difference (MID) Based on EORTC QLQ-C30 and EORTC QLQ-EN24

| Subscale | Individual Items | MID | Deterioration from<br>Baseline |
|---|---|---|---|
| EORTC QLQ-C30 Functional scales | | | the appli |
| Physical functioning | 1-5 | 6 | Decrease (CFB ≤ -MID) |
| Role functioning | 6-7 | 7 subject | Decrease (CFB $\leq$ -MID) |
| Emotional functioning | 21-24 | 7 5110, | Decrease (CFB $\leq$ -MID) |
| Cognitive functioning | 20, 25 | 40 | Decrease (CFB $\leq$ -MID) |
| Social functioning | 26-27 | 6 | Decrease (CFB $\leq$ -MID) |
| Global health status | 26-27<br>29-30 | | |
| Quality of life | 29-30 | 5 and 10 | Decrease (CFB $\leq$ -MID) |
| Symptom scales/items | | | |
| Fatigue | 10, 12, 18 | 6 | Increase (CFB $\geq$ MID) |
| Nausea and vomiting | 14-15 | 4 | Increase (CFB $\geq$ MID) |
| Pain | 9, 19 | 7 | Increase (CFB $\geq$ MID) |
| Dyspnoea | 8 | 5 | Increase (CFB $\geq$ MID) |
| Insomnia | 11 | 5 | Increase (CFB $\geq$ MID) |
| Appetite loss | 13 | 6 | Increase (CFB $\geq$ MID) |
| Constipation | 16 | 6 | Increase (CFB $\geq$ MID) |
| Diarrhoea | 17 | 4 | Increase (CFB $\geq$ MID) |
| Financial difficulties | 28 | 4 | Increase (CFB $\geq$ MID) |
| EORTC QLQ-EN24 | | | |
| Functional scales | | | |
| Sexual interest | 49 | 5 | Decrease (CFB $\leq$ -MID) |
| Sexual activity | 50 | 5 | Decrease (CFB $\leq$ -MID) |

Table 7.b Definition of Minimally Important Difference (MID) Based on EORTC QLQ-C30 and EORTC QLQ-EN24

| Subscale | Individual Items | MID | Deterioration from Baseline |
|---|---|---|---|
| Sexual enjoyment | 54 | 5 | Decrease (CFB ≤-MID) |
| Symptom scales | | | licar |
| Lymphoedema | 31-32 | 5 | Increase (CFB $\geq$ MID) |
| Urological symptoms | 34-37 | 5 | Increase (CFB $\geq$ MID) |
| Gastrointestinal symptoms | 38-42 | 5 | Increase (CFB $\geq$ MID) |
| Poor body image | 47-48 | 5 | Increase (CFB $\geq$ MID) |
| Sexual/vaginal problems | 51-53 | 5 | Increase (CFB $\geq$ MID) |
| Pain in back and pelvis | 33 | 5, 5 | Increase (CFB $\geq$ MID) |
| Tingling/numbness | 43 | 3 | Increase (CFB $\geq$ MID) |
| Muscular pain | 44 | 5 | Increase (CFB $\geq$ MID) |
| Hair loss | 45 | 5 | Increase (CFB $\geq$ MID) |
| Taste change | 46 | 5 | Increase (CFB $\geq$ MID) |

Note: CFB = change from baseline.

Differences between treatment groups in the EORTC QLQ-C30 subscales, the global health status/QOL score and EORTC QLQ-EN24 subscales will be evaluated using published minimally important difference (MID) as shown in Table 7.2. At each visit up to cycle 12 and by treatment, present the number and percentage of patients for each of the following categories for each subscale scores:

- Worsened: EORTC QLQ-C30 functional scores, global health status/QOL score, EORTC QLQ-EN24 score : change from baseline ≤ -MID, for symptom scores: change from baseline ≥ MID
- Improved: EORTC QLQ-C30 functional scores, global health status/QOL score, EORTC QLQ-EN24 score: change from baseline ≥ MID, symptom scores: change from baseline ≤ MID.
- Stable: change from baseline within MID.

In addition, at each visit and by treatment, the cumulative number and cumulative percentage whose change from baseline of the subscale scores reflects improvement will be summarized.

### 7.10.3 Time to Deterioration

Time to deterioration is defined as the time from the date of randomization to the date of first detection of deterioration for each EORTC QLQ-C30 subscales, the global health status/QOL score, and for each EORTC QLQ-EN24 score [date of first detection of deterioration – date of randomization + 1]. Deterioration is defined as a change from baseline  $\geq$  MID for EORTC QLQ-C30 symptom scores and as a change from baseline  $\leq$  -MID for EORTC QLQ-C30 function scores, global health status/QOL score and EORTC QLQ-EN24 score (see Table 7.2). Patients without deterioration will be censored at their last quality of life assessment. For patients with no post-baseline assessment, time to deterioration will be censored at Day 1.

The Kaplan-Meier method will be used to analyze the distribution of time to deterioration for each treatment arm. Kaplan-Meier survival curves, the 25th, 50th (median), and 75th percentiles, along with associated 2-sided 95% confidence intervals (CIs), hazard ratio estimated using Cox regression model with treatment arm and stratification factors as covariates along with associated 95% CI for comparison of paclitaxel to paclitaxel+MLN0128, paclitaxel to MLN0128 and paclitaxel to MLN0128+MLN1117, and Kaplan-Meier estimates at 6, 12, 18 and 24 months will be presented. A stratified log-rank test will be performed to compare the time to deterioration between treatment arms. The stratification factors are the histological subtype (endometrioid vs. non-endometrioid), the lines of prior chemotherapy (1 vs. 2) and prior taxane therapy (yes vs. no). The original IRT stratification factors will be used in models.

### 7.11 Safety Analysis

All safety analyses will be performed using the Safety population.

### 7.11.1 Adverse Events

Toxicity will be evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 4.03, effective date 14 June 2010.

Treatment-emergent AEs that occur after administration of the first dose of study drug and through 30 days after the last dose of study drug will be tabulated.

Tabular summaries by MedDRA system organ class and preferred term will be provided for the following:

- Treatment-emergent adverse events.
- Drug-related TEAEs.
- Grade 3 or higher TEAEs.
- Grade 3 or higher drug-related TEAEs.
- Most commonly reported TEAEs (at least 10% in any arm, sorted by preferred term).
- Serious adverse events.
- Most frequent non-serious TEAEs (> 5% in any arm).

Patients reporting the same event more than once will have that event counted only once within each system organ class, and once within each preferred term.

Adverse events of interest will be tabulated for the following:

| Adverse event of interest | MedDRA Preferred Term | |
|---|---|---|
| Asthenic Conditions | Asthenia, Decreased activity, Fatigue, Malaise, Sluggishness (modified HLT) | |
| Mucosal Inflammation | Enanthema | Allergic stomatitis |
| | Mucosa vesicle | Aphthous ulcer |
| | Mucosal atrophy | Lip erosion |
| | Mucosal discolouration | Lip ulceration |
| | Mucosal dryness | Mouth ulceration |
| | Mucosal erosion | Oral mucosa erosion |
| | Mucosal exfoliation | Palatal ulcer |
| | Mucosal haemorrhage | Stomatitis |
| | Mucosal hyperaemia | Stomatitis haemorrhagic |
| | Mucosal hypertrophy | Stomatitis necrotising |
| | Mucosal induration | |
| | Mucosal inflammation | |
| | Mucosal membrane<br>hyperplasia | |
| ,0 | Mucosal necrosis | |
| * akedai. For no | Mucosal pain | |
| · . | Mucosal pigmentation | |
| Teore | Mucosal roughness | |
| ( \Q_{II} | Mucosal toxicity | |
| O | Mucosal ulceration | |
| | Mucous membrane disorder | |
| | Oedema mucosal | |
| | Mucosal infection | |

| Adverse event of interest | MedDRA Preferred Term |
|---|---|
| | Mucosal excoriation |
| | Erythroplasia |
| | Burning sensation mucosal |
| | Burning sensation mucosal Paraesthesia mucosal Leukoplakia Drug eruption Fixed eruption Mucocutaneous haemorrhage Mucocutaneous rash |
| | Leukoplakia |
| | Drug eruption |
| | Fixed eruption |
| | Mucocutaneous haemorrhage |
| Rash | Mucocutaneous naemorrhage Mucocutaneous rash Nodular rash Rash Rash Rash erythematous Rash generalised Rash macular Rash maculo-papular Rash maculovesicular Rash morbilliform Rash papular Rash rubelliform Rash scarlatiniform Rash vesicular |

# 7.11.1.1 Deaths

All deaths occurring on-study and during follow-up will be displayed (regardless of treatment-emergent AE status). On-study death is defined as death that occurs between the first dose of study drug and 30 days after the last dose of study drug (adverse events with an outcome of death).

All cause mortality will be tabulated, which includes death of all causes, deaths related to disease under study, and deaths due to other reasons. On-study deaths will be tabulated, which includes deaths related to disease under study, deaths due to other reasons, and deaths within 30 and 60 days of first dose.

### 7.11.1.2 Clinical Laboratory Evaluations

Whenever available, laboratory values will be assigned toxicity grades using the NCI CTCAE version 4.03. The number and proportion of patients with shifts in NCI CTCAE toxicity grades from baseline to the worst post baseline toxicity grade will be summarized for the following laboratory tests:

- Hematology: Hemoglobin increased, Activated partial thromboplastin time (aPTT)
  prolonged, INR increased, Lymphocyte count decreased, Lymphocyte count increased,
  Neutrophil count decreased, Platelet count decreased, White blood cell count decreased
- Chemistry: Alanine aminotransferase (ALT) increased, Alkaline phosphatase increased,
  Aspartate aminotransferase (AST) increased, Bilirubin (total) increased, Cholesterol high,
  Creatinine increased, Gamma glutamyl transferase (GGT) increased, Corrected Calcium decreased, Corrected Calcium increased, Glucose decreased, Glucose increased,
  Potassium decreased, Potassium increased, Magnesium decreased, Magnesium increased, Sodium decreased, Sodium increased, Triglycerides increased, Albumin decreased, Phosphate decreased, Amylase increased

The shift from baseline to worst post baseline will include scheduled and unscheduled visits.

For fasting glucose, the shifts from baseline to the worse post baseline (2 hours only) will be summarized for MLN0128 QW and MLN0128 + MLN1117 arms.

The actual values (in SI units) and change from baseline in clinical laboratory parameters will be summarized by treatment group for Neutrophils (ANC), Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Glucose, Hemoglobin A1c, Cholesterol (total), Triglycerides, High-density lipoprotein cholesterol (HDL-C) and Low-density lipoprotein cholesterol (LDL-C) up to 12 cycles. Figures of mean actual values over time will also be generated for these clinical laboratory parameters (in SI units).

## 7.11.2 Vital Signs

The actual values and change from baseline for vital sign parameters including temperature, heart rate, systolic and diastolic blood pressure, and weight, will be summarized over time for each treatment arm up to 6 cycles.

### 7.11.3 12-Lead ECGs

The actual values and change from baseline for ECG results (QT, QTcF, PR interval, QRS interval, Ventricular Rate) will be summarized over time for each treatment group up to 6 cycles. In addition, the number and percent of patients with increases >30 ms and >60 ms from pre-dose in QTcF will also be summarized over time up to 6 cycles.

All QT values will be converted to QTcF using Fridericia's correction:

$$QT_F = \frac{QT}{\sqrt[3]{RR}}_{\text{(sec)}}$$

Shifts from baseline to the worst post-baseline ECOG score will be tabulated by treatment arm up to 6 cycles.

7.12 Interim Analysis

As specified in 41.

### As specified in the protocol

There will be 2 interim analyses with early stopping rules for futility in both the single-agent MLN0128 and MLN0128 + MLN1117 arms using the Bayesian predictive probability design. The endpoint for the interim analysis will be based on the number of patients who achieve complete or partial response of any duration, or stable disease  $\geq 16$  weeks as assessed by the investigator (clinical benefit at 16 weeks). The decision rule for the interim analyses is derived based on the following assumptions:

- Ineffective CBR-16 rate (Ho): 30%.
- Effective CBR-16 rate (Ha): 50%.
- Alpha = 10%; power = 80%.
- Prior Beta Distribution Parameters:  $\alpha_0 = 0.30$ ,  $\beta_0 = 0.70$ .
- The probability of early termination under the null hypothesis is 77%.

Each interim analysis will be based on patients who have had the opportunity to complete a minimum of 4 cycles or have discontinued study drug before the end of Cycle 4. The data cut-off is when the 20<sup>th</sup> patient achieves end of Cycle 4 in the treatment arms single-agent MLN0128 and MLN0128 + MLN1117. For all patients, use data up to Cycle 4 for interim analysis. Based on the first 20 patients in each arm, 1 or both arms may be dropped if at most 6 patients experience clinical benefit at 16 weeks in each arm. After the first 30 patients in each arm have been evaluated following 4 cycles of treatment, 1 or both arms may be dropped if at most 10 patients experience clinical benefit at 16 weeks in each arm.

For the interim analysis CBR at 16 weeks is defined as the number of patients who achieve CR or PR at the end of cycle 2 or end of cycle 4, or have SD at the end of Cycle 2 and at the end of Cycle 4 (based on unconfirmed response.).

### Futility analysis

An additional futility analysis will be performed when 50% of PFS events have occurred for the paclitaxel and paclitaxel+MLN0128 treatment arms. The decision rule is based on a Bayesian framework: posterior probability (true HR > **0.78** | observed HR) is greater than 70%. The futility criteria will be met if the observed PFS HR for the comparison of paclitaxel vs paclitaxel+MLN0128 at the interim analysis for futility is greater than or equal to 0.898.

- 1. QOL instruments, EORTC QLQ-C30 and EORTC QLQ EN24, will be analyzed over time
- 2. The Per-protocol population was added to the analysis populations.
- QOL instruments, EORTC QLQ-C30 and EORTC QLQ EN24, will be analyzed over time and not restricted to just change from baseline to end of study visit as stated in the protocol. The Per-protocol population was added to the analysis populations.

  For PFS analysis, patients who started alternate subsequent therapy prior to disprogression will be censored at the date of last adsubsequent therapy. The progression will be consored at the date of last adsubsequent therapy. 3. For PFS analysis, patients who started alternate subsequent therapy prior to disease subsequent therapy. The protocol did not explicitly state this condition.
- 4. In addition to Kaplan-Meier method that will be used to analyze distribution of PFS, OS and TTP for each treatment arm and the p-values from a stratified log-rank test, the HRs and 95% CIs from a stratified Cox regression model with treatment arm and stratification factors as covariates will also be presented for comparison of paclitaxel to paclitaxel+MLN0128, paclitaxel to MLN0128 and paclitaxel to MLN0128+MLN1117. The protocol did not explicitly state the model for estimating the HRs.
- 5. The secondary endpoints e.g. ORR, CBR, CBR-16 and DOR will be based on both confirmed and unconfirmed best overall response.
- property of Takedai. For non-commercial use 6. Added details for the sensitivity analyses based on IRC review of scans. The IRC will only be performed for Arms A (paclitaxel) and B (paclitaxel + MLN0128).

Probeth of Takeda: For non-commercial use only and subject to the applicable Terms of Use

In addition to the analysis outputs outlined above in the main text, separate by-patient listings will also be generated to include the following information:

• Disposition of subjects.

• Demographic and other baseline characteristics (including stratification factors)

• Important protocol deviations (including flag to in the per protocol.

- Hand subject to the from the per protocol population).
- Concomitant medications.
- Follow-up anti-cancer therapy.
- TEAEs resulting in discontinuation of study drug.
- SAEs.
- Deaths and cause of death.
- Sparse PK data.
- RECIST response assessment and best overall response based on investigator assessment and IRC assessment [Arms A (paclitaxel) and B (paclitaxel + MLN0128) only].

## **Appendix B: Date Imputation Rules**

### Incomplete Dates in the Screening Period

- 1. If only the day-component is missing, the first day of the month will be used if the year and the month are the same as those for the first dose of study drug. Otherwise, the fifteenth will be used.
- 2. If only the year is present, and it is the same as the year of the first dose of study drug, the fifteenth of January will be used unless it is later than the first dose, in which case the date of the first of January will be used.
- 3. If only the year is present, and it is not the same as the year of the first dose of study drug, the fifteenth of June will be used.

# Incomplete Adverse Event Onset Date

Assumption: For on-study Adverse Events.

If *year* is missing (or completely missing): set to the date of first dose.

If (year is present and month and day are missing) or (year and day are present and month is missing):

If *year* = year of first dose: set the date to the first dose date.

If *year* < year of first dose: set *month* and *day* to December 31<sub>st</sub>.

If *year* > year of first dose: set *month* and *day* to January 1st.

If *month* and *year* are present and *day* is missing:

If year = year of first dose, and:

If *month* = month of first dose: set *day* to day of first dose.

If *month* < month of first dose: set *day* to last day of *month*.

If *month* > month of first dose: set *day* to 1st day of *month*.

If *year* < year of first dose: set *day* to last day of month.

If *year* > year of first dose: set *day* to 1st day of month.

For all other cases: set to date of first dose.

### Incomplete Concomitant Medication Start Date

If *year* is missing (or completely missing): do not impute.

applicable Terms of Use applicable terms If (year is present and month and day are missing) or (year and day are present and month id subject to is missing):

Set month and day to January 1st.

If *year* and *month* are present and *day* is missing:

Set day to 1st day of month.

### Incomplete Concomitant Medication End Date

If *year* is missing (or completely missing): do not impute.

If (year is present and month and day are missing) or (year and day are present and month is missing):

Set month and day to December 31st.

If *year* and *month* are present and *day* is missing:

Set day to last day of the month.

## Incomplete Subsequent Anti-Cancer Therapy Start Date

If year is missing (or completely missing): set to date of last dose of study treatment + 1 If (year is present and month and day are missing) or (year and day are present and month is missing):

If year > year of the last dose: Set month and day to January 1st.

If year = year of the last dose: Set *month* and *day* to date of last dose of study

treatment +1

If year and month are present and day is missing:

Set day to 1st day of month if the resulting imputed date is greater than date of last

Otherwise set the imputed date to date of last dose + 1

# ELECTRONIC SIGNATURES

| | Signed by | Meaning of Signature | Server Date (dd-MMM-yyyy HH;mm 'UTC') |
|---|---|---|---|
| PPD | | Biostatistics Approval | 07-Sep-2018 20:06 UTC |
| | | Clinical Science Approval | 07-Sep-2018 20:08 UTC |
| | | Biostatistics Approval | 07-Sep-2018 21:23 UTC |
| | | iole | |
| | | Meaning of Signature Biostatistics Approval Clinical Science Approval Biostatistics Approval ercital use only and subjections are also also and subjections are also and subjections are also and subjections are also and subjections are also | |
| | | ercialuse | |
| | of Non-comi | | |
| 79 | Eggi. Ko. | | |
| property of ' | | | |